CLINICAL TRIAL: NCT01766024
Title: International Multicenter Randomized Double-blind Crossover Study of Pharmacokinetics, Pharmacodynamics and Tolerability of BCD-033 (CJSC BIOCAD, Russia) and Rebif® (Merck Serono S.p.А., Italy) After Single Subcutaneous Administration to Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics Study of BCD-033 Compared to Rebif® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-033-1
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: interferon beta-1a; pharmacokinetics; pharmacodynamics; volunteers
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-033 → Rebif (Experimental): Volunteers in this group initially will receive a single sc injection of the study drug BCD-033 (interferon beta-1a) at a dose of 44 µg (on Day 1) and then, after at least 14 days, a single sc injection of the reference drug Rebif® (interferon beta-1a) at a dose of 44 µg.
  Interventions: Drug: Interferon beta-1a
- Rebif → BCD-033 (Experimental): Volunteers in this group initially will receive a single sc injection of active comparator Rebif (interferon beta-1a) at a dose of 44 µg (on Day 1) and then, after at least 14 days, a single sc injection of the study drug BCD-033 (interferon beta-1a) at a dose of 44 µg.
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Interferon beta-1a — Each volunteer will receive 1 subcutaneous (sc) injection of the study drug BCD-033 (interferon beta-1a) and 1 sc injection of active comparator Rebif (interferon beta-1a) at a dose of 44 µg with an interval of at least 14 days.
  Other Names: BCD-033; Rebif

SUMMARY:
This is a randomized double-blind crossover study of pharmacokinetics, pharmacodynamics and tolerability of BCD-033 (interferon beta-1a manufactured by CJSC BIOCAD, Russia) and Rebif® (Merck Serono S.p.A.., Italy) in healthy volunteers. The purpose of the study is to demonstrate the non-inferiority of pharmacokinetics, pharmacodynamics and tolerability parameters after single subcutaneous injection. Each dtug will be administered to each volunteer at a dose of 44 µg as a single subcutaneous injection with an interval of at least 14 days.

DETAILED DESCRIPTION:
Each dtug (BCD-033 and Rebif) will be administered to each volunteer at a dose of 44 µg as a single subcutaneous injection with an interval of at least 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Male gender;
* Age 18 - 45 years inclusive;
* Body mass index (BMI) (18,5 - 24,99 kg/m2);
* Healthy condition proven by the volunteer's history, global assessment and laboratory analysis results:
* Absence in past medical history and at screening of clinically significant dysfunctions of circulatory, respiratory, nervous, hematopoietic, endocrine and digestive systems, liver and kidneys;
* Haematology and biochemistry tests, urinalysis and thyroid hormone analysis results are within normal limits according to standards of the study site. Screening laboratory analyses should be performed not more than 14 days before volunteer's inclusion in the study;
* Hemodynamic parameters are within normal limits: systolic blood pressure - from 100 to 139 mmHg, diastolic blood pressure - from 60 to 90 mmHg, heart rate - from 50 to 90 bpm;
* Absence of history of chronic infection (tuberculosis) and chronic inflammation;
* Absence of HIV, hepatitis B and C virus, syphilis;
* Absence of acute infections within 4 weeks before inclusion in the study;
* Absence of psychiatric disorders and other conditions that can interfere with volunteer's ability to follow the study protocol, including depression;
* Well-being (in volunteer's opinion) within 30 days before participation in the study;
* Absence of history of systematic alcohol and drug abuse;
* Ability of the volunteer, in investigator's opinion, to follow the study protocol procedures and requirements;
* Willingness of volunteers and their sexual partners of childbearing potential to use reliable contraception methods starting from 2 weeks before inclusion into the study and until 4 weeks after receiving the last dose of the investigational products. This criterion is not applicable to patients who underwent surgical sterilization. Reliable contraceptive measures include one barrier method in combination with one of the following methods: spermicides, intrauterine device or oral contraceptives used by participant's partner;
* Consent to avoid alcohol intake within 24 hours before and 8 days after each administration of the test or reference drugs;
* Consent to avoid grapefruit juice (or other products containing grapefruit) intake within 72 hours before and 8 days after each administration of the study or reference drugs.

Exclusion Criteria:

* Previous use of IFN-β1-containing medications at any time before inclusion;
* History of serious allergic reactions (anaphylaxis or multiple allergy);
* Known allergy or intolerance to interferons or any other components of study or reference drugs;
* Major surgery within 30 days before screening;
* Impossibility to install venous catheter for blood sampling (e.g. because of skin disorders at the sites of venipuncture);
* Diseases or other conditions that can interfere with the investigational drugs pharmacokinetics (e.g. chronic liver, kidney, blood, circulatory system, lung or neuroendocrine diseases, including diabetes mellitus and others);
* History of epileptic seizures;
* Regular oral or parenteral use of any medications including over-the-counter drugs, vitamins and nutritional additives within less than 2 weeks before inclusion in the study;
* Intake of medications, including over-the-counter drugs and biologically active additives that can influence hemodynamics, liver function etc. (barbiturates, omeprazole, cimetidine etc.) within less than 30 days before inclusion in the study;
* Intake of medications that influence immune status (cytokines and their inductors, glucocorticoids etc.) within less than 30 days before participation in the study;
* Smoking more than 10 cigarettes per day;
* Subjects who consume more than 10 units of alcohol per week or who have history of alcohol abuse or evidence of drug/chemical abuse (one unit of alcohol equals ½ l [500 ml] of beer, one glass [200 ml] of wine or l shot glass [50 ml] of spirits);
* Donation of 450 ml and more of blood or plasma within 2 months before inclusion in the study;
* Participation in other clinical studies within less than 1 month before inclusion in the study or simultaneous participation in another clinical study;
* Previous participation in this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Sardaryan, PhD, Principal Investigator — City Mariin Hospital
Locations (1):
- City Mariin Hospital, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCD-033 → Rebif | Rebif → BCD-033
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-033 → Rebif | Rebif → BCD-033 | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Area Under Concentration-time Curve (AUC) of Interferon (IFN) Beta-1a From the Moment of Drug Administration Until 48 Hours and to Infinity(AUC(0-48) and AUC(0-∞) Respectively)
Description: Primary outcome measure for pharmacokinetics analysis. Blood samples were taken before the injection, then after 15 min, 30 min, 45 min, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours and 48 hours.
Time Frame: 0 to 48 hours post-dose
Measure: Median (Inter-Quartile Range); unit: (pg/ml)•h
Groups:
- BCD-033: the endpoint was assessed in all the volunteer who received BCD-033
- Rebif: the endpoint was assessed in all the volunteer who received Rebif
Arm/Group | BCD-033 | Rebif
Number analyzed (Participants) | 30 | 30
(pg/ml)•h | 6318.3 [5368.4 to 7484.9] | 6807.9 [5714.9 to 8920.1]

2. Primary Outcome: Cmax of Interferon Beta-1a
Description: Primary outcome measure for pharmacokinetics analysis Blood samples were taken before the injection, then after 15 min, 30 min, 45 min, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours and 48 hours.
Time Frame: 0 to 48 hours post-dose
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- BCD-033: the endpoint was assessed in all the volunteer who received BCD-033 (interferon beta-1a)
- Rebif: the endpoint was assessed in all the volunteer who received Rebif (interferon beta-1a) a
Arm/Group | BCD-033 | Rebif
Number analyzed (Participants) | 30 | 30
pg/ml | 104.9 [80.2 to 123.4] | 102.4 [83.6 to 148.6]

3. Primary Outcome: AUC(0-168) and AUC(0-∞) of Neopterin and MxA Protein
Description: Primary outcome measure for pharmacodynamics analysis. Blood samples were taken before the injection, then after 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours.
Time Frame: 0 to 168 hours post-dose
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*h
Arm/Group | BCD-033 | Rebif
Number analyzed (Participants) | 32 | 32
(ng/ml)*h
  neopterin | 552.7 [458.1 to 661.6] | 537.6 [392.6 to 680.1]
  MxA protein | 2444.2 [2005.5 to 3011.2] | 2131.2 [1728.0 to 3245.0]

4. Secondary Outcome: Тmax of Interferon Beta-1a Blood Samples Were Taken Before the Injection, Then After 15 Min, 30 Min, 45 Min, 1 Hour, 2 Hours, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours and 48 Hours.
Description: Secondary outcome measure for pharmacokinetics analysis
Time Frame: 0 to 48 hours post-dose
Reporting Status: Not Posted

5. Secondary Outcome: Т½ of Interferon Beta-1a Blood Samples Were Taken Before the Injection, Then After 15 Min, 30 Min, 45 Min, 1 Hour, 2 Hours, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours and 48 Hours.
Description: Secondary outcome measure for pharmacokinetics analysis
Time Frame: 0 to 48 hours post-dose
Reporting Status: Not Posted

6. Secondary Outcome: Кel of Interferon Beta-1a Blood Samples Were Taken Before the Injection, Then After 15 Min, 30 Min, 45 Min, 1 Hour, 2 Hours, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours and 48 Hours.
Description: Secondary outcome measure for pharmacokinetics analysis
Time Frame: 0 to 48 hours post-dose
Reporting Status: Not Posted

7. Secondary Outcome: Cl of Interferon Beta-1a Blood Samples Were Taken Before the Injection, Then After 15 Min, 30 Min, 45 Min, 1 Hour, 2 Hours, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours and 48 Hours.
Description: Secondary outcome measure for pharmacokinetics analysis
Time Frame: 0 to 48 hours post-dose
Reporting Status: Not Posted

8. Secondary Outcome: Cmax of Neopterin and MxA Protein Blood Samples Were Taken Before the Injection, Then After 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 Hours.
Description: Secondary outcome measure for pharmacodynamics analysis
Time Frame: 0 to 168 hours post-dose
Reporting Status: Not Posted

9. Secondary Outcome: Tmax of Neopterin and MxA Protein
Description: Secondary outcome measure for pharmacodynamics analysis
Time Frame: 0 to 168 hours post-dose
Reporting Status: Not Posted

10. Secondary Outcome: Adverse Event (AE) and Serious Adverse Event (SAE) Incidence
Description: Secondary outcome measure for safety assessment
Time Frame: up to Day 43
Reporting Status: Not Posted

11. Secondary Outcome: AE of Garde 3-4 Incidence
Description: Secondary outcome measure for safety assessment
Time Frame: up to Day 43
Reporting Status: Not Posted

12. Secondary Outcome: Local Reaction Incidence
Description: Secondary outcome measure for tolerability assessment
Time Frame: up to Day 43
Reporting Status: Not Posted

13. Secondary Outcome: Study Withdrawal Rate Due to AE
Description: Secondary outcome measure for safety assessment
Time Frame: up to Day 43
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | BCD-033 | Rebif
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 32/32 | 32/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-033 (N=32) | Rebif (N=32)
Flu-like syndrom (General disorders) | 32 (32) | 32 (32) — Fever, aches, chills, headache, weakness
Local reactions (General disorders) | 13 (13) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other